CLINICAL TRIAL: NCT03223129
Title: Insulin Sensitivity and Metabolomics During Oral Administration of Glucose and a Graded Intravenous Infusion in Patients With Normal Glucose Tolerance, Impaired Glucose Tolerance and in Patients With Type 2 Diabetes Mellitus
Brief Title: Insulin Sensitivity and Metabolomics During Oral Administration of Glucose and Graded Intravenous Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: U911/14
Record Dates: First submitted 2017-06-12; First posted 2017-07-19 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Impaired glucose tolerance; Metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Patients with either normal glucose tolerance, impaired glucose tolerance or with diagnosed type 2 diabetes mellitus will undergo oral glucose tolerance tests with an increasing load of glucose and thereafter isoglycemic intravenous glucose infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with normal glucose tolerance (Other): Patients included in this arm will have a plasma glucose below 140 mg/dl after a 2 h oral glucose tolerance test with a glucose load of 75 g.
  All patients in this arm will undergo oral glucose tolerance test with increasing glucose load and a graded intravenous glucose infusion were plasma glucose levels are held at the same level as during the oral glucose tolerance test.
  Interventions: Other: Oral glucose tolerance test; Other: Graded intravenous glucose infusion
- Patients with impaired glucose tolerance (Other): Patients included in this arm will have a plasma glucose between 140 mg/dl to 199 mg/dl after a 2 h oral glucose tolerance test with a glucose load of 75 g.
  All patients in this arm will undergo oral glucose tolerance test with increasing glucose load and a graded intravenous glucose infusion were plasma glucose levels are held at the same level as during the oral glucose tolerance test.
  Interventions: Other: Oral glucose tolerance test; Other: Graded intravenous glucose infusion
- Patients with type 2 diabetes mellitus (Other): Patients included in this arm will have a plasma glucose above 200 mg/dl after a 2 h oral glucose tolerance test with a glucose load of 75 g.
  All patients in this arm will undergo oral glucose tolerance test with increasing glucose load and a graded intravenous glucose infusion were plasma glucose levels are held at the same level as during the oral glucose tolerance test.
  Interventions: Other: Oral glucose tolerance test; Other: Graded intravenous glucose infusion

INTERVENTIONS:
Other: Oral glucose tolerance test — Oral glucose tolerance tests were glucose is administrated orally with an increasing load (25g, 75g, 100 g)
Other: Graded intravenous glucose infusion — Graded intravenous glucose infusion where glucose is infused in order to receive an plasma glucose pattern comparable to those received during the oral glucose tolerance tests.

SUMMARY:
Bariatric surgery has been proven to be an effective treatment of type 2 diabetes and it has highlighted to role of the small intestine in glucose homeostasis. Improvement of glucose homeostasis occurs just a few days after the bariatric surgery, where parts of the small intestine is bypassed, has been performed. Furthermore, conditioned medium from the duodenum and the jejunum from both diabetic rodents and humans are able to induce insulin resistance in normal mice and in myocytes. Hence the hypothesis is that the small intestine secretes factors that are able to induce insulin resistance.

This project aims to study how orally ingested glucose is able to induce insulin resistance and if this response differs in patients with normal glucose tolerance, impaired glucose tolerance and in patients with type 2 diabetes mellitus. To address this question glucose homeostasis will be studied by comparing whole body glucose uptake during a progressively increased oral glucose load with a graded glucose infusion where the blood glucose levels will be kept in the same range as during the oral glucose load in patients with normal glucose tolerance, impaired glucose tolerance and patients with type 2 diabetes mellitus.

Previous studied have shown that different metabolites and bile acids could be involved the regulation of glucose homeostasis. Hence, it is possible that the gut regulates metabolites that could be involved in small intestine-induced insulin resistance described above. The aim of this research is to study metabolomics in plasma collected during the oral glucose tolerance test with increasing load of glucose and the graded glucose infusion where plasma glucose level will be held in the same levels as during the oral glucose tolerance test and study the differences in patients with normal glucose tolerance, impaired glucose tolerance and in patients with type 2 diabetes mellitus.

The expected results in this study will demonstrate that the gut plays an important role in glucose homeostasis and that this system is dysregulated in type 2 diabetes. More importantly, novel factors derived or regulated from the gut that regulate insulin resistance and glucose tolerance will be identified which could be possible targets for future antidiabetic therapies.

DETAILED DESCRIPTION:
The incidence of obesity and obesity-associated metabolic disorders such as insulin resistance and type 2 diabetes is increasing worldwide. To date, bariatric surgery is the only obesity treatment that results in long-term weight reduction. In addition, bariatric surgery has been reported to promote remission of type 2 diabetes and to be a more effective treatment than standard medication for type 2 diabetes. Surprisingly, improvement in glucose homeostasis after some bariatric surgery procedures occurs before weight loss is achieved. The mechanisms behind this improvement are still unclear but a recent study indicates that the bypassing of jejunum could play an important role in glucose homeostasis. Moreover, jejunum-derived proteins present in serum in both human and mice induce insulin resistance in cell cultures of myocytes and in mice. This taken together indicates that the gut may play an important role in glucose homeostasis in type 2 diabetes mellitus.

Metabolomics has recently been regarded to be one of the most suitable technologies for investigating complex diseases such as type 2 diabetes mellitus because it represent a real-time functional portrait of the organisms. Previous studies have shown that different metabolites and bile acids could be involved in the regulation of glucose homeostasis. Hence it is possible that the gut regulates metabolites that could be involved in the impaired glucose tolerance and type 2 diabetes mellitus.

The specific aims of this research project are:

Aim 1: To demonstrate that orally ingested glucose induces insulin resistance and to determine if this regulation of glucose homeostasis differs between subjects with normal glucose tolerance, impaired glucose tolerance and subjects with type 2 diabetes mellitus.

Aim 2: To identify metabolites regulated by the gut that are associated with impaired glucose tolerance and type 2 diabetes mellitus.

To address this aim, differences in glucose kinetics will be studied when glucose is orally administrated (in an oral glucose tolerance test, OGTT) compared to an graded intravenous glucose infusion, were plasma glucose levels are held in the same range as during the OGTT, in subjects with normal glucose tolerance (n = 8), impaired glucose tolerance (n = 8) and type 2 diabetes mellitus (n = 8).

Basal glucose kinetics will first be assessed by double glucose tracer technique. In the basal part of the glucose tolerance tests glucose tracer nr 1 will be infused and then be followed by either a continued infusion and a gradually increasing oral glucose load (25 g, 75 g and 125 g with a 2 h interval during the OGTT) with glucose tracer nr 2 or an graded intravenous glucose tracer infusion where plasma glucose levels are adjusted to those obtained during the OGTTs.

Gas chromatography/mass spectrometry will be used to measure isotopic enrichment of glucose tracers. Insulin, glucagon, total glucagon-like peptide 1 (GLP-1) and C-peptide will be measured by radioimmunoassays repeatedly during the glucose tolerance tests. Glucose kinetics including endogenous glucose production, insulin sensitivity and insulin secretion will be calculated. Differences in glucose kinetics between the oral and intravenous administration of glucose will be calculated and compared in subjects with normal glucose tolerance, impaired glucose tolerance or type 2 diabetes mellitus.

Analysis of metabolomics will be performed in plasma collected during the OGTT and the graded intravenous glucose infusion. Metabolites in plasma samples will be analyzed using two global profiling analytical platforms and a targeted profiling platform. Two-dimensional gas chromatography coupled to time-of-flight mass spectrometry (GCxGC-TOFMS) will be performed to measure small polar metabolites. Molecular lipids will be assessed by a global platform using ultra performance liquid chromatography coupled to quadrupole-TOFMS (UPLC-QTOFMS). A targeted platform based on UPLC coupled to triple-quadrupole MS (UPLC-QqQMS) will be performed to quantify both unconjugated and conjugated forms of bile acids.

Differences in plasma metabolites during OGTT and graded intravenous glucose infusion will be studied to assess information on possible regulation by the gut and the results will be compared in subjects with normal glucose tolerance, impaired glucose tolerance and subjects with type 2 diabetes mellitus.

Significance The expected results in this study will demonstrate that the gut plays an important role in glucose homeostasis and that this system is dysregulated in type 2 diabetes. More importantly, novel factors derived or regulated from the gut that regulate insulin resistance and glucose tolerance will be identified which could be possible targets for future antidiabetic therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65
* BMI between 35 and 60 kg/m2
* Ability to understand and comply with the study process.

Exclusion Criteria:

* History of type 1 diabetes or secondary diabetes;
* Previous bariatric surgery;
* History of medical problems such as mental impairment;
* Major cardiovascular disease;
* Major gastrointestinal disease;
* Major respiratory disease;
* Hormonal disorders;
* Infection;
* History of drug addiction and/or alcohol abuse;
* Internal malignancy;
* Pregnancy;
* Suspected or confirmed poor compliance;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Glucose kinetics | 1 year
  Whole body glucose uptake will be measured using a double glucose tracer technique during both the oral glucose tolerance test and the graded intravenous glucose infusion.

SECONDARY OUTCOMES:
Metabolomics | 1 year
  Plasma levels of small polar metabolites, molecular lipids and conjugated and unconjugated bile acids will be measured during both oral glucose tolerance test and during the graded intravenous glucose infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD PhD, Principal Investigator — The Catholic University of the Sacred Heart
Locations (1):
- Università Cattolica S. Cuore, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mingrone G, Panunzi S, De Gaetano A, Ahlin S, Spuntarelli V, Bondia-Pons I, Barbieri C, Capristo E, Gastaldelli A, Nolan JJ. Insulin sensitivity depends on the route of glucose administration. Diabetologia. 2020 Jul;63(7):1382-1395. doi: 10.1007/s00125-020-05157-w. Epub 2020 May 8. PMID 32385603